CLINICAL TRIAL: NCT01917760
Title: The Pharmacokinetics of Gamma-aminobutyric Acid in Healthy Volunteers.
Brief Title: Pharmacokinetics Study of Gamma-aminobutyric Acid
Acronym: GABA-PK
Status: Completed | Type: Observational
Sponsor: Huashan Hospital (Other)
Collaborators: Unity Health Toronto (Other); University of Florida (Other); University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Zhaoyun Zhang, professor of endocrinology and metabolism, Huashan Hospital
Other Study IDs: KY-2013-222; JDRF_17-2013-499 (Registry Identifier: Juvenile Diabetes Research Foundation International (JDRF)])
Record Dates: First submitted 2013-07-06; First posted 2013-08-07 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Diabetes Mellitus; Diabetes Mellitus, Type 1; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases; Autoimmune Diseases; Immune System Diseases
Keywords: Gamma-aminobutyric acid; Pharmacokinetics; Pharmacodynamics; Insulin; C-peptide; Glucagon
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases; Autoimmune Diseases; Immune System Diseases; Insulin Resistance

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — This is an open-labeled, 3-phase, self-control study. In phase 1, blood is sampled from volunteers who will take placebo to obtain the baseline value. In phase 2, volunteers will take a single oral dose of 2000 mg GABA. There are at least 7 days between the two phases. In phase 3, volunteers will take a repeated oral dose of 2000 mg GABA (thrice daily for seven days). There are at least 5-7 days between phase 3 and phase 3. In each phase, individuals will be observed for 24 hours to obtain the complete concentration time curve. 4 ml of blood will be sampled at the following time-point for predose and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 and 24 hour postdose.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine upon administering GABA orally to a person how it is absorbed, distributed, as well as the drug's pharmacological effects on the body such as glucose levels, serum C-peptide and/or insulin levels (referred to as pharmacokinetics/pharmacodynamics). We will conduct experiments in normal subjects to address these questions.

DETAILED DESCRIPTION:
Type 1 diabetes is an autoimmune disease resulting from the progressive loss of pancreatic insulin-secreting beta-cells. This consequently leads to a lack of insulin and elevation of blood sugar, namely hyperglycemia, which is a major cause for the development of diabetes and its acute or chronic complications. The current treatment for type 1 diabetes requires a life-long dependency on daily insulin injections, causing inconvenience and burden to patients. Drug-induced hypoglycemia is also common as it presents a major challenge in insulin therapy. Furthermore, although insulin therapy is lifesaving, it is not a cure as it neither reverses the progression of the disease nor prevents the development of serious complications associated with this disease. New treatments are urgently needed.

Recent studies have demonstrated that a natural chemical found in the brain, gamma-aminobutyric acid (GABA), which is also produced in large quantities by pancreatic beta-cells, has beta-cell regenerative and immunoregulatory effects. Importantly, GABA prevented and partially reversed diabetes in type 1 diabetes mouse models. It is important to address essential questions regarding the potential effects of GABA in diabetic patients in humans. Given the largely unknown mechanism of action of GABA in the pancreas, and the limited information on how GABA is absorbed, distributed and eliminated from the human body, we plan to examine these issues (referred to as pharmacokinetics/pharmacodynamics) in normal subjects.

The outcome of this study will provide useful information on the mechanism of action of GABA in human subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteers in good health condition between 19 and 40 years of age (inclusive) at the time of signing the informed consent.
2. Body mass index (BMI) between 18.5 and 24 kg/m2 (inclusive), with weight greater than 50 kg.
3. Not on any medication 2 weeks before screening.
4. No blood donation within 3 months before screening.
5. Must sign the informed consent. Note: Blood and biochemical tests must be normal during the screening. However, if the participant's test-results were beyond the normal range, the individual can still be recruited as long as the results do not affect the experiment.

Exclusion Criteria:

1. Abnormalities of physical examination, laboratory tests, or ECG in screening, which may influence the results of the study.
2. Previous or existing history of severe heart, liver, kidney, gastrointestinal, nervous system, mental, or metabolic abnormalities as well as other diseases which can affect drug absorption, circulation, metabolism, or excretion.
3. History of alcoholism, smoking, or drug abuse within the past 1 year.
4. Participation in any clinical drug study within the past 30 days.
5. Any definite or suspected allergy or family history of allergy to GABA or any other similar drugs.

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Residents of Shanghai
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2013-07; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
pharmacokinetic characteristics of γ-aminobutyric acid (GABA) | baseline and up to 30 days
  The primary endpoint of this study is to obtain the pharmacokinetic characteristics of γ-aminobutyric acid (GABA), including:
  1. Area under the plasma concentration-time curve from time 0 to the last quantifiable concentration (AUC0-t),
  2. Area under the plasma concentration-time curve from time 0 extrapolated to infinity (AUC0-∞),
  3. Maximum observed plasma concentration (Cmax),
  4. Time to maximum plasma concentration (Tmax), and
  5. Terminal elimination half-life in plasma (t½)

SECONDARY OUTCOMES:
serological characteristics | baseline and up to 30 days
  plasma glucose levels, insulin, C-peptide and glucagon levels will be measured

OTHER OUTCOMES:
Exploratory measures | baseline and up to 30 days
  plasma glucagon-like peptide-1 (GLP-1) and glycated serum protein (GSP)will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Yiming Li, Principal Investigator — Huashan Hospital; Qinghua Wang, Principal Investigator — Huashan Hospital/St Michael's Hospital; Zheng Jiao, Principal Investigator — Huashan Hospital
Locations (1):
- Department of Endocrinology and Metabolism，Huashan hospital, Shanghai, Shanghai Municipality, China